CLINICAL TRIAL: NCT04236089
Title: Compare Effects of the Mirror Therapy and Robotic Mirror Therapy in Electroencephalography of Healthy Adults and Stroke Patients.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201900537A3
Record Dates: First submitted 2020-01-17; First posted 2020-01-22 (Actual); Last update posted 2021-03-04 (Actual); Status verified 2020-01

CONDITIONS: Healthy Adults; Stroke Patients
Keywords: mirror therapy; robotic mirror therapy; Electroencephalography; stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- mirror therapy of healthy adults (No Intervention): Traditional mirror therapy in electroencephalography of healthy adults.
- robotic mirror therapy of healthy adults (Experimental): Robotic mirror therapy in electroencephalography of healthy adults.
  Interventions: Device: robotic hand
- mirror therapy of stroke patients (No Intervention): Traditional mirror therapy in electroencephalography of stroke patients.
- robotic mirror therapy of stroke patients (Experimental): Robotic mirror therapy in electroencephalography of stroke patients.
  Interventions: Device: robotic hand

INTERVENTIONS:
Device: robotic hand — mirror therapy with robotic hand
  Arms: robotic mirror therapy of healthy adults; robotic mirror therapy of stroke patients

SUMMARY:
Mirror therapy has recently attracted increasing attention; however, most patients have the difficulties to perform mirror therapy due to limited imaginary ability. A mirror robotic hand system was developed, which consisted with a wearable exoskeletal hand, sensor glove, and a control box. The patient's unaffected hand wears the sensor glove, the affected hand wears the wearable exoskeleton hand, and the unaffected hand does the certain transitive and intransitive tasks as the mirror group, and then makes the affected hand do the same movements driven by the exoskeleton robotic hand. The investigators hypothesize that combining both approaches might facilitate the sensorimotor cortex that controls movement and might augment somatosensory input and further treatment efficacy. This study is aimed at investigating the effects of Mirror therapy and robotic mirror therapy on motor cortical activations in healthy adults and stroke patients using electroencephalography. All participants will perform the conditions of resting, moving right hand with or without robotic hand as the baseline data, then they will do mirror therapy using the right hand as active hand, or wearing robotic hand doing mirror therapy in random sequence. Electroencephalography (EEG) assessment will be done to assess the neurophysiologic effects of the different interventions. The investigators will use a questionnaire to assess the subjective opinion about the different interventions.

combined with execution (video AOE). The investigators will use the pair-t test to assess the within subjects differences in EEG and the questionnaire results.

This study will be done during 2020/02/01 - 2021/03/31.

ELIGIBILITY:
Inclusion Criteria:

* healthy adults: right handed, with normal upper extremity and cognition functions
* stroke patients:one side upper limb spasticity

Exclusion Criteria:

* 1. wrist weakness or deformity 2. skin problem 3. musculoskeletal injury of upper extremities

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Electroencephalography assessment | 1.5hours
  Compare the brainwave of the different interventions through Fourier Transform

SECONDARY OUTCOMES:
Questionnaire | 30 minutes
  Collect the subjective opinion about the different interventions

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Rehabilitation, Chang Gung Memorial Hospital-Kaohsiung Medical Center, Kaohsiung, Taiwan, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No